CLINICAL TRIAL: NCT05178966
Title: Evaluation of the Effectiveness of a Day Patient-caregiver Psychoeducationnal Program on the Burden of Caregivers
Brief Title: Evaluation of Efficiency of One Day Patient/Caregiver Psychoeducation on the Caregiver's Burden
Acronym: BP ONEDAY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-A01317-34; 2021-A01317-34 (Other: ANSM)
Record Dates: First submitted 2021-09-24; First posted 2022-01-05 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Bipolar Disorder; Caregiver Burden
Keywords: bipolar disorder; psychoeducation; caregivers; burden; stigmatization
MeSH Terms: conditions — Bipolar Disorder; Caregiver Burden; Stereotyping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bp OneDay programm (Experimental): The BP One-Day program is based on a single day of psychoeducation .
  Interventions: Behavioral: Bp OneDay psychoeducation program
- Waiting List (No Intervention): Patients assigned in control group will be placed in waiting list and will benefit from the program after their participation to this study. During study participation, they will receive treatment as usual.

INTERVENTIONS:
Behavioral: Bp OneDay psychoeducation program — The BP One-Day Psychoeducation program is based on a single day of psychoeducation . This program was carried out by members of the bipolar expert center network in various hospitals of the network and included :
  * Representation of BD
  * Definition, diagnosis and awareness of the disorder
  * Depressive, hypo / manic symptoms
  * Vulnerability to BD causes of BD, risk factors for relapses
  * Drug treatments, drug compliance and non-drug treatments
  * Early detection of prodromal signs
  * Communication techniques
  Each BP One-Day psychoeducation session welcomes an average of ten participants (5 patients / 5 caregivers). At the end of the day, participants receive a booklet containing the main information of the day.
  BP One-Day program is delivered by a nurse and a psychologist specialized in both BD and therapy group facilitation. A specialized psychiatrist intervenes in the section "Medication treatments and medication adherence" for a period of approximately one hour.
  Arms: Bp OneDay programm

SUMMARY:
Bipolar disorder (BD) has a huge impact on the lives of patient and their relatives. Psychoeducation programs on BD has been shown to be effective on the burden of patients and their caregivers. However, actual programs appear to be incompatible with patients obligations and services requirements of the service. The development of "minute" programs (in one day) is justified.

DETAILED DESCRIPTION:
Bipolar disorder (BD) has a huge impact on patient lives and their relatives. BD psychoeducation has been shown to be effective on patient disease course and caregivers burden. However, the programs offered appear to be incompatible with the participants obligations and services requirements. In this context we wanted to develop a "minute" program (Bp one day).

Study participation includes 3 visits : inclusion visit and 2 follow up visits.

The main objective is to assess the effectiveness of day psychoeducational program (BP OneDay) on caregiver burden at one month according to the Zarit Caregiver Burden Interview (ZCBI) total score.

This study also aims to assess the effectiveness of BP OneDay on caregiver stigma, patient self-stigma and medication adherence, quality of life, and bipolar disorder knowledge.

The study is an open-label randomized controlled trial with two arms

Overall, 120 dyads will be recruited randomly affected in 2 groups :

* the interventional group will benefit from a day psychoeducational program : Bp oneDay
* the control group will be placed on the waiting list

The benefits expected from Bp OneDay are to reduce caregiver burden and stigma and improve knowledge about BD. For patients, we expect improve disease understanding, drug adherence and reduce self-stigmatization. If the results are promising, this program can be widely disseminated and thus increase cares' solution for patients and relatives in large urban centers.

ELIGIBILITY:
Patient inclusion Criteria:

* Be over 18 years old;
* Meet the criteria for bipolar disorder (I, II, unspecified) according to the DSM-5 criteria;
* Be able to understand the nature, purpose and methodology of the study;
* Presence of a caregiver

Patient Exclusion Criteria:

* Subject unable to adhere to the group requirements (cognitive disorder, decompensated mood state ...);
* Subject protected by law (subject under guardianship and / or guardianship) or deprived of liberty by a judicial or administrative decision;
* Subject unable to understand, speak and write French;
* Subject in a period of exclusion from another protocol.
* Subject not having signed an informed consent
* Subject not affiliated with a social security scheme or such a scheme

Caregiver inclusion criteria ;

* Subject over 18 years old;
* Subject designated as a regular caregiver of a patient with bipolar disorder. A regular caregiver is a trusted person designated by the patient as being one of his main support, having knowledge of the diagnosis of bipolar disorder and who can be called upon in the context of care.
* Subject able to understand the nature, purpose and methodology of the study;

Caregiver exclusion criteria :

* Subject unable to adhere to the groupre quirements (cognitive disorder, decompensated mood state ...);
* Subject protected by law (subject under guardianship and / or curatorship) or deprived of liberty by a judicial or administrative decision ;
* Subject unable to understand, speak and write French;
* Subject in a period of exclusion from another protocol.
* Subject not having signed an informed consent
* Subject not affiliated with a social security scheme or such a scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
caregivers burden | Day65 for experimental group, Day35 for control group
  evaluation of caregiver burden based on the Zarit Caregiver Burden Interview total score.
  The Zarit Caregiver Burden Interview is a self-administered questionnaire assessing caregiver burden using 22 items. Five themes are examined: psychological and physical suffering, financial, relational and social difficulties. For each of the 22 items, the caregiver determines how often he feels a given emotion in the helping relationship. This frequency ranges from 0 "never" to 4 "Almost always". The overall score is obtained by adding all the items together, it varies from 0 to 88. The higher the score, the greater the burden felt by the caregiver.

SECONDARY OUTCOMES:
caregivers stigmatization | Day44 for experimental group, Day14 for control group
  évaluation of caregivers stigmatization using Affiliate stigma scale on caregivers of people with mental illness The Affiliate stigma scale on caregivers of people with mental illness is a self-questionnaire composed of 22 items assessing 3 dimensions of stigma : the cognitive, affective and behavioral dimension. Participants are asked to rate their level of agreement with the statements on a 4-point Likert scale (ranging from 1 "Strongly disagree" to 4 "Strongly agree). The total score ranges from 22 to 88. The higher the score, the more severe the stigma.
caregivers stigmatization | Day65 for experimental group, Day35 for control group
  évaluation of caregivers stigmatization using Affiliate stigma scale on caregivers of people with mental illness The Affiliate stigma scale on caregivers of people with mental illness is a self-questionnaire composed of 22 items assessing 3 dimensions of stigma : the cognitive, affective and behavioral dimension. Participants are asked to rate their level of agreement with the statements on a 4-point Likert scale (ranging from 1 "Strongly disagree" to 4 "Strongly agree). The total score ranges from 22 to 88. The higher the score, the more severe the stigma.
Internalized Stigma of patients | Day44 for experimental group, Day14 for control group
  evaluation of Internalized Stigma according to the Internalized Stigma of Mental Illness total score This self-questionnaire consists of 29 items. Each item is rated using a 4-points Likert scale ranging from 1 "Strongly disagree" to 4 "Strongly agree". The 29 items are grouped according to 5 themes: alienation (the fact of not feeling a full member of the society in which we live), approval of stereotypes, perceived discrimination, social withdrawal, and resistance to stigma. The higher the score, the more severe the self-stigma.
Internalized Stigma of patients | Day65 for experimental group, Day35 for control group
  evaluation of Internalized Stigma according to the Internalized Stigma of Mental Illness total score This self-questionnaire consists of 29 items. Each item is rated using a 4-points Likert scale ranging from 1 "Strongly disagree" to 4 "Strongly agree". The 29 items are grouped according to 5 themes: alienation (the fact of not feeling a full member of the society in which we live), approval of stereotypes, perceived discrimination, social withdrawal, and resistance to stigma. The higher the score, the more severe the self-stigma.
Patient quality of life | Day44 for experimental group, Day14 for control group
  Evaluation of patient quality of life according to the Quality of Life Enjoyment and Satisfaction Questionnaire Short Form total score.
  This 16-items self-administered questionnaire assesses the quality of life through the assessment of physical health, social relationships, family relationships, mood, libido, the ability to function on a daily basis, the ability to invest and enjoy leisure time, to work, the economic level, the place of life and the general feeling of well-being. The last two items assess satisfaction with treatment as well as satisfaction with life and are treated independently of the others. Each item is scored on a 5-point Likert scale and represents the level of satisfaction experienced over the last week. A calculation of the overall score is performed for items 1 to 14 (ranging from 14 to 70) and is expressed as a percentage (0-100). The higher the score, the better the quality of life.
Patient quality of life | Day65 for experimental group, Day35 for control group
  Evaluation of patient quality of life according to the Quality of Life Enjoyment and Satisfaction Questionnaire Short Form total score.
  This 16-items self-administered questionnaire assesses the quality of life through the assessment of physical health, social relationships, family relationships, mood, libido, the ability to function on a daily basis, the ability to invest and enjoy leisure time, to work, the economic level, the place of life and the general feeling of well-being. The last two items assess satisfaction with treatment as well as satisfaction with life and are treated independently of the others. Each item is scored on a 5-point Likert scale and represents the level of satisfaction experienced over the last week. A calculation of the overall score is performed for items 1 to 14 (ranging from 14 to 70) and is expressed as a percentage (0-100). The higher the score, the better the quality of life.
caregivers quality of life | Day44 for experimental group, Day14 for control group
  Evaluation of caregivers quality of life according to the Quality of Life Enjoyment and Satisfaction Questionnaire Short Form total score.
  This 16-items self-administered questionnaire assesses the quality of life through the assessment of physical health, social relationships, family relationships, mood, libido, the ability to function on a daily basis, the ability to invest and enjoy leisure time, to work, the economic level, the place of life and the general feeling of well-being. The last two items assess satisfaction with treatment as well as satisfaction with life and are treated independently of the others. Each item is scored on a 5-point Likert scale and represents the level of satisfaction experienced over the last week. A calculation of the overall score is performed for items 1 to 14 (ranging from 14 to 70) and is expressed as a percentage (0-100). The higher the score, the better the quality of life.
caregivers quality of life | Day65 for experimental group, Day35 for control group
  Evaluation of caregivers quality of life according to the Quality of Life Enjoyment and Satisfaction Questionnaire Short Form total score.
  This 16-items self-administered questionnaire assesses the quality of life through the assessment of physical health, social relationships, family relationships, mood, libido, the ability to function on a daily basis, the ability to invest and enjoy leisure time, to work, the economic level, the place of life and the general feeling of well-being. The last two items assess satisfaction with treatment as well as satisfaction with life and are treated independently of the others. Each item is scored on a 5-point Likert scale and represents the level of satisfaction experienced over the last week. A calculation of the overall score is performed for items 1 to 14 (ranging from 14 to 70) and is expressed as a percentage (0-100). The higher the score, the better the quality of life.
Medication Adherence | Day44 for experimental group, Day14 for control group
  Evaluation of patient medication adherence according to Medication Adherence Rating Scale total score.
  This self-questionnaire has 10 yes / no items. The total score varies between 0 and 10. The higher the score, the better the compliance. This scale was created and is widely used in the psychiatric population.
Medication Adherence | Day65 for experimental group, Day35 for control group
  Evaluation of patient medication adherence according to Medication Adherence Rating Scale total score.
  This self-questionnaire has 10 yes / no items. The total score varies between 0 and 10. The higher the score, the better the compliance. This scale was created and is widely used in the psychiatric population.
Bipolar disorder Knowledge in patients | Day44 for experimental group, Day14 for control group
  Evaluation of Bipolar Disorde knowledge in patients according to "Quizz BP" total score.
  This self-administered questionnaire is composed of twenty true or false questions. It addresses different themes: occurrence, etiology, semiology, factors triggering episodes, comorbidities, treatments. The overall score fluctuates between 0 and 20. Although this test has not been validated, it has already been used in several published works
Bipolar disorder Knowledge in patients | Day65 for experimental group, Day35 for control group
  Evaluation of Bipolar Disorde knowledge in patients according to "Quizz BP" total score.
  This self-administered questionnaire is composed of twenty true or false questions. It addresses different themes: occurrence, etiology, semiology, factors triggering episodes, comorbidities, treatments. The overall score fluctuates between 0 and 20. Although this test has not been validated, it has already been used in several published works
Bipolar disorder Knowledge in caregivers | Day44 for experimental group, Day14 for control group
  Evaluation of Bipolar Disorde knowledge in caregivers according to "Quizz BP" total score.
  This self-administered questionnaire is composed of twenty true or false questions. It addresses different themes: occurrence, etiology, semiology, factors triggering episodes, comorbidities, treatments. The overall score fluctuates between 0 and 20. Although this test has not been validated, it has already been used in several published works
Bipolar disorder Knowledge in caregivers | Day65 for experimental group, Day35 for control group
  Evaluation of Bipolar Disorde knowledge in caregivers according to "Quizz BP" total score.
  This self-administered questionnaire is composed of twenty true or false questions. It addresses different themes: occurrence, etiology, semiology, factors triggering episodes, comorbidities, treatments. The overall score fluctuates between 0 and 20. Although this test has not been validated, it has already been used in several published works
Patient satisfaction | Day44 for experimental group, Day14 for control group
  Evaluation of patient satisfaction with the group according to a liker score ranged from 0 "absolutely not satisfied" to 10 "Extremely satisfied"
caregiver satisfaction | Day44 for experimental group, Day14 for control group
  Evaluation of caregiver satisfaction with the group according to a liker score ranged from 0 "absolutely not satisfied" to 10 "Extremely satisfied"

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Montpellier, Montpellier, France